CLINICAL TRIAL: NCT05423548
Title: Analysis of Risk Factors of Neurodevelopmental Disorder in Deaf Infants Under Ten Months of Age.
Acronym: EnTNDre
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220048
Record Dates: First submitted 2022-02-17; First posted 2022-06-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Congenital Sensorineural Hearing Loss
Keywords: Congenital sensorineural hearing loss; Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with congenital deafness: Children with congenital deafness followed in the ENT department of the Necker hospital and having benefited before their 10 months, from a pilot consultation, filmed, jointly carried out by a child psychiatrist from the Therapeutic Childhood and Deafness Unit of St Maurice Hospitals (UTES) and a psychologist from the ENT department of Necker for the neurodevelopmental risk assessment, between May 2018 to April 2020.

SUMMARY:
Among risk factors of neurodevelopmental disorder is congenital hearing loss. However, congenital deafness is neither necessary nor sufficient for the occurrence of warning signs of neurodevelopmental disorder. The investigative team hypothesizes that the co-occurrence of these two clinical entities results from a common origin, within a syndromic diagnosis including other medical issues. These situations would therefore be very different from those of babies suffering from isolated sensorineural deafness.

This study aims to identify which factors are statistically correlated with the association of congenital deafness and early symptoms of neurodevelopmental disorder, thanks to a partnership between a regional center for psychiatry of deaf children (Therapeutic Childhood and Deafness Unit of St Maurice Hospitals, UTES) and a pediatric audiophonology department (ENT department of the Necker-Enfants Malades hospital).

This work is based on a cohort of 26 children under ten months of age diagnosed with severe to profound congenital sensorineural hearing loss. As part of their pre-implantation cochlear assessment, a consultation was filmed to precisely analyze the interactional and sensorimotor skills of these children (clinical observations, administration of a specific evaluation grid called Olliac Grid), after reviewing the films. The investigative team will then be able to grade the neurodevelopmental risk.

In order to clarify what factors are linked with a neurodevelopmental risk, medical data concerning the child's family context, birth, and audiological profile will also be collected, and put in perspective with the assessed neurodevelopmental risk gradation.

DETAILED DESCRIPTION:
Congenital deafness remains among well-known risk factors for Neurodevelopmental Disorders, in particular Autism Spectrum Disorders (ASD). According to current data of the literature, the risk of ASD in children with hearing loss is twice as high as in the general population. Furthermore, while the main aim of French government strategy for autism 2018-2022 is to promote early detection and intervention, it is noted that deaf children suffer from a significant diagnostic delay with regard to autism spectrum disorders.

Today it is possible to detect clinical warning signs of a neurodevelopmental impairment since the first months of life. The investigative team believe that these warning signs present a risk for further severe disability such as ASD, Attention Deficit / Hyperactivity Disorder (ADHD), learning disorders and so on, that is to say every psychiatric diagnosis included in neurodevelopmental disorders as the DSM-V classifies them. This encourages clinicians to assess every new-born with high risk factors of neurodevelopmental disorder.

No research has been conducted on the screening of Autism Spectrum Disorders (and more broadly of Neurodevelopmental Disorders) in deaf infants and the correlations with their clinical profile (health conditions, psychomotor development and typology of deafness).

One of the difficulties lies in the fact that these children constitute a heterogeneous population. Studying deaf infants requires taking into account multiple parameters, such as etiology of the hearing loss, associated disorders, or early life history. Moreover, first months of a born-deaf child are a highly emotional and demanding period for parents. However, the investigative team hope that observing this population will help better understand what constitutes in newborns with congenital hearing loss, associated risk factors for autism.

Knowing that congenital deafness is neither necessary nor sufficient for the early occurrence of a neurodevelopmental warning signs, the investigative team hypothesizes that the co-occurrence of these two medical conditions results from a common origin, as a syndromic diagnosis including other medical issues. These situations would therefore be very different from those of babies suffering from isolated sensorineural deafness.

The investigative team aim to identify which factors are statistically correlated with the association of congenital deafness and early diagnosis of clinical signs of neurodevelopmental risk, thanks to a partnership between a regional center for psychiatry of deaf children (Therapeutic Childhood and Deafness Unit of St Maurice Hospitals, UTES) and an infant audiophonology department (ENT department of the Necker-Enfants Malades hospital).

This work is based on a cohort of 26 infants under ten months of age diagnosed with severe to profound congenital sensorineural hearing loss. The enrollment of the patients took place from May 2018 to April 2020, based on consultations for the management of deafness in the audiophonology department of the Necker Enfants Malades Hospital in Paris.

As part of the pre-implantation cochlear assessment carried out in the audiophonology department of the Necker Enfants Malades Hospital, each child in the cohort has attended a consultation to assess the risk of neurodevelopmental disorder. This pilot consultation was carried out by a child psychiatrist from the UTES together with a psychologist from the ENT department of Necker, and was filmed to precisely analyze the interactional skills of the children (clinical observations, administration of a specific evaluation grid called Olliac Grid (Olliac et al, 2017), gradation of the neurodevelopmental risk), after reviewing the films.

Anamnesis data concerning the family context (parental and sibling history) and birth (antenatal conditions, term, per and post-natal complications) will be collected, with particular attention to the elements already identified in the literature as associated with risk of Neurodevelopmental Disorders. In order to clarify what factors are linked with a neurodevelopmental risk, medical data concerning the child's family context, birth, and audiological profile will be collected, and put in perspective with the previously assessed neurodevelopmental risk gradation.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital deafness
* Follow-ups in the ENT department of the Necker hospital
* Having benefited from a pilot consultation, filmed, jointly carried out by a child psychiatrist from Therapeutic Childhood and Deafness Unit of St Maurice Hospitals (UTES) and a psychologist from the Necker ENT department for the assessment of neurodevelopmental risk
* Pilot consultation carried out before the child is 10 months old
* Information of the holders of parental authority and collection of their non-opposition to the study

Exclusion Criteria:

* Children assessed after 10 months
* Opposition of legal representatives for the use of their child's medical data and of the film

Max Age: 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with congenital deafness followed in the ENT department of the Necker hospital and having benefited before their 10 months, from a pilot consultation, filmed, jointly carried out by a child psychiatrist from the Therapeutic Childhood and Deafness Unit of St Maurice Hospitals Therapeutic Childhood and Deafness Unit of St Maurice Hospitals (UTES) and a psychologist from the ENT department of Necker for the neurodevelopmental risk assessment.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Children's interactional behaviours | 12 months
  From the study of the psychiatric assessment filmed, children will be seprated in 2 categories wether they present interactional warning signs of neurodevelopmental disorders (NDD) or not.
  The children's interactional behaviours quality will be assessed using the Olliac grid : a standardized clinical assessment of an infant's ability to initiate an interaction and/or respond to one (Olliac et al, 2017). According to answers to 4 questions about an infant's behaviors during a health appointment, a score will be attributed. The maximum score is 15 and means good ability to interact with parents and unknown people. A score ≤ 3 or ≤ 5, depending on the infant's age is considered "at risk" for autism spectrum disorder (ASD).
  Children will be considered presenting Interactional Warning Signs of NDD if they have an " at risk " score at the Olliac grid, which means a total score ≤ 3 for children aged between 4 months and 8 months + 30 days, and a score ≤ 5 for children aged over 9 months.
Warning signs of neurodevelopmental disorders | 12 months
  From the study and the description of the psychiatric assessment carried out and filmed, children will be seprated in two descriptive categories wether they present warning signs of neurodevelopmental disorders or not.
  The sensorimotor development of children will be described from the video recording and compared to the development of a typical hearing child.
  Children will be considered presenting sensorimotor warning signs of NDD if they exhibit two or more of the following conditions:
  * Global hypertonia or hypotonia
  * Jolt in response to visual, tactile, or vestibular moderate stimuli
  * Repetitive dorsal hyperextensions
  * Motor restlessness
  * Lack of motor fluidity
  * Excessive use of thoraco-pneumatic tonus
  * Motor development delay These conditions are known to reflect psychomotor development vulnerability, and are easy to assess by experienced early childhood professionals.

SECONDARY OUTCOMES:
Perinatal complication | 12 months
  Description of clinical profiles of the children from medical file. Comparison of frequencies of perinatal complication between infants presenting warning signs of NDD and infants who don't. The clinical data will be compared in terms of percentages, following a binary measure (present/absent).
  Any perinatal complication will count for "present". Here is some examples of what could be considered : premature delivery threat, fetal growth restriction, gestational diabetes, emergency ceasarean section, low birth weight, neonatal resuscitation, hyperbilirubinemia.
Preterm birth | 12 months
  Description of clinical profiles of the children from medical file. Preterm birth is a major cause of NDD. This clinical data will be compared in terms of percentages, following a binary measure (present/absent) between infants presenting warning signs of NDD and infants who don't.
  Comparison of frequencies of preterm birth. Any birth under 37 weeks of gestation will be counted as "present".
Neonatal positive Cytomegalovirus (CMV) status | 12 months
  Description of clinical profiles of the children from medical file. Neonatal positive Cytomegalovirus (CMV) status is a major cause of congenital hearing loss, and a risk factor of NDD. This clinical data will be compared in terms of percentages, following a binary measure (present/absent) between infants presenting warning signs of NDD and infants who don't. A positive CMV status will be considered as "present".
Sensorimotor disturbances in the first months | 12 months
  Description of clinical profiles of the children from medical file. The clinical data will be compared in terms of percentages, following a binary measure (present/absent) between infants presenting warning signs of NDD and infants who don't.
  Comparison of frequencies of causes of sensorimotor disturbances in the first months: any of the following conditions will be counted as "present": gastrostomy, feeding disorder, and/or Gastroesophageal reflux.
Vestibular hyporeflexia or areflexia | 12 months
  Description of clinical profiles of the children from medical file. The clinical data will be compared in terms of percentages, following a binary measure (present/absent) between infants presenting warning signs of NDD and infants who don't.
  Comparison of frequencies of vestibular dysfunction. Either vestibular hyporeflexia or areflexia will be considered as "present". These data are available in every audiophonologic medical file, as every deaf infant gets a vestibular assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Loundon, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Salomé Akrich, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akrich S, Parlato de Oliveira E, Favrot-Meunier C, Rebichon C, de Clerck A, Ettori S, Rouillon I, Prang I, Loundon N. Analysis of specific risk factors of neurodevelopmental disorder in hearing-impaired infants under ten months of age: "EnTNDre" an opening research stemming from a transdisciplinary partnership. Int J Pediatr Otorhinolaryngol. 2023 Mar;166:111453. doi: 10.1016/j.ijporl.2023.111453. Epub 2023 Jan 21. PMID 36746056